CLINICAL TRIAL: NCT01250184
Title: Treatment of Myofascial Pain Syndrome With Lidocaine Injection and Physical Therapy, Alone or in Combination: a Single-blind, Randomized, Controlled Clinical Trial.
Brief Title: Treatment of Myofascial Pain Syndrome With Lidocaine Injection and Physical Therapy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo Rehabilitacion en Salud (Network)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Luz Helena Lugo Agudelo, Associate Professor, Grupo Rehabilitacion en Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrupoRS0001
Record Dates: First submitted 2010-11-27; First posted 2010-11-30 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Myofascial Pain Syndrome; Pain; Myofascial Trigger Point Pain; Musculoskeletal Pain
Keywords: Myofascial pain; Trigger points.; Lidocaine injection.; Physical therapy
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain; Musculoskeletal Pain | interventions — Physical Therapy Modalities; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical Therapy (Active Comparator): Twelve sessions, 3 per week.
  Interventions: Other: Physical therapy
- Lidocaine injection (Active Comparator): Blocking the myofascial trigger point (MTP) with lidocaine injection, unique dose.
  Interventions: Drug: Lidocaine injection
- Lidocaine injection + physical therapy (Experimental): Blocking the Myofascial trigger point (MTP) with lidocaine injection plus a standarized therapeutic exercise program, twelve sessions, 3 per week.
  Interventions: Other: Lidocaine injection + physical therapy

INTERVENTIONS:
Other: Physical therapy — Twelve sessions (3 per week)
  Other Names: standardized therapeutic exercise program
  Arms: Physical Therapy
Drug: Lidocaine injection — blocking the Myofascial trigger point (MTP) with lidocaine injection, unique dose.
  Other Names: blocking the Myofascial trigger point
  Arms: Lidocaine injection
Other: Lidocaine injection + physical therapy — blocking the Myofascial trigger point (MTP) with lidocaine injection plus a standarized therapeutic exercise program (twelve sessions, 3 per week)
  Other Names: blocking plus a standarized therapeutic exercise program
  Arms: Lidocaine injection + physical therapy

SUMMARY:
Background: Myofascial pain syndrome (MPS) of the shoulder girdle and cervical region is a common musculoskeletal problem that is often chronic or recurrent. It has demonstrated the effectiveness of different treatments such as exercise, injection but not comparing them with each other. The objective of this research was to demonstrate whether lidocaine injection into trigger points combined with a physical therapy program was more effective than each separatetreatment in improving pain, function and quality of life in a group of patients with myofascial pain syndrome (MPS) of the shoulder girdle and cervical region.

Design: Single-blind, randomized, controlled clinical trial with three parallel groups in the departments of physical medicine and rehabilitation of two urban hospitals. There were 127 patients with myofascial pain in the shoulder girdle for more than six weeks in length and pain greater than 40 mm on the visual analog scale (VAS). There were three intervention groups: physical therapy (PT), lidocaine injection (LI), or the combination of both (PT + LI). The primary outcome at one month was the VAS, and the secondary outcomes were measured using the SF36 pain scaleat one and three months.

Keywords: Myofascial pain, trigger points, lidocaine injection, physical therapy.

DETAILED DESCRIPTION:
We propose a double blind randomized controlled clinical trial, in different health centers in Medellin. The subjects are patients with myofascial trigger points (MTP) in muscles of the shoulder girdle (levator scapulae, trapezius, infraspinatus) diagnosed by neck ans shoulder pain lasting langer than 6 weeks, and that have not received rehabilitation treatment and are not currently taking analgesic medications. We have calculated a sample of 45 patients in each group.

The physical and rehabilitation doctors who evaluated the patients and the nurse who assessed the patients were blinded to treatment allocation. Physicians who performed the MTP injection did not participate in the evaluation of primary and secondary outcomes. Physical therapists who conducted the therapeutic exercise program did not participate in the evaluation of primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Cervical Pain at least six weeks
* At least 40 mm in the VAS
* They cannot been received treatment like physical therapy or analgesics
* Maximum score of PHQ 16 points

Exclusion Criteria:

* Depression
* Fibromyalgia
* Cervical Radiculopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luz H Lugo Agudelo, Professor, Principal Investigator — Universidad de Antioquia Grupo Rehabilitacion en Salud
Locations (2):
- Colombia (2):
  - Clinica de Las Américas, Medellín, Antioquia
  - Ips Universitaria, Medellín, Antioquia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the databases of two general and specialized medical institutions, 762 patients were identified to have non-specific myalgia or muscle disorders diagnoses. A nurse by phone and two medical physiatrists at the hospitals, with over 10 years of research experience evaluated the MPS patients and their medical history.
Pre-assignment Details: The randomization process was performed using permuted blocks.This process was performed by an investigator (HIG) who had no contact with the patients. The allocations to each treatment were placed in consecutive sealed, opaque envelopes, were kept in the research headquarters and were taken to the site according to the number of patients referred.
Groups:
- Lidocaine Injection + Physical Therapy: Blocking the Myofascial trigger point (MTP) with lidocaine injection plus a standarized therapeutic exercise program, twelve sessions, 3 per week.
  blocking the MTP plus physical therapy: blocking the Myofascial trigger point (MTP) with lidocaine injection plus a standarized therapeutic exercise program (twelve sessions, 3 per week)
- Lidocaine Injection: Blocking the myofascial trigger point (MTP) with lidocaine injection, unique dose.
  Blocking the MTP: blocking the Myofascial trigger point (MTP) with lidocaine injection, unique dose.
Period: Overall Study
Arm/Group | Physical Therapy | Lidocaine Injection + Physical Therapy | Lidocaine Injection
Started | 43 | 41 | 43
Completed | 43 | 41 | 43
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was calculated with the software "Sample Size Javeriana University" it was took in to account a error type I of 0.05, type II of 0.2, number of measurements before randomization = 1, after performing the randomization = 2, correlation between measurements of 0.6, clinically important difference of 0.35, for a number of patients = 45 each
Groups:
- Blocking the MTP Plus Physical Therapy: Blocking the Myofascial trigger point (MTP) with lidocaine injection plus a standarized therapeutic exercise program, twelve sessions, 3 per week.
  blocking the MTP plus physical therapy: blocking the Myofascial trigger point (MTP) with lidocaine injection plus a standarized therapeutic exercise program (twelve sessions, 3 per week)
- Blocking the MTP: Blocking the myofascial trigger point (MTP) with lidocaine injection, unique dose.
  Blocking the MTP: blocking the Myofascial trigger point (MTP) with lidocaine injection, unique dose.
- Total: Total of all reporting groups
Arm/Group | Blocking the MTP Plus Physical Therapy | Physical Therapy | Blocking the MTP | Total
Number analyzed (Participants) | 41 | 43 | 43 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (11.1) | 42.6 (9.7) | 37.7 (11.8) | 39.19 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 33 | 104
  Male | 6 | 7 | 10 | 23
Region of Enrollment [Number; unit: participants]
  Colombia | 41 | 43 | 43 | 127
Concomitant factors [Number; unit: participants] — A patient could have more than one Concomitant factor
  participants
    Stress | 34 | 29 | 30 | 93
    Sleeplessness | 24 | 18 | 23 | 65
    Longer positions | 27 | 34 | 29 | 90
Muscles with trigger point [Number; unit: participants] — A patient could have more than one trigger point
  participants
    Trapezius muscle | 37 | 42 | 39 | 118
    Levator scapulae | 31 | 27 | 26 | 84
    Infraspinatus muscle | 12 | 12 | 13 | 37
Physical examination [Number; unit: participants] — A patient could have more than one alteration on the physical examination.
  participants
    Sensitive Alteration | 8 | 7 | 8 | 23
    Referred pain | 22 | 36 | 23 | 81
    Local twitch response | 29 | 26 | 22 | 77
Visual Analogue Scale for Pain [Mean (Standard Deviation); unit: units on a scale] — VAS with a score of 0-100, where 100 is the value representing the highest degree of pain and 0 the lowest. Successful treatment was defined as a reduction in pain of at least 20% of the previous score on the VAS after 4 weeks of the initial evaluation, or 14 mm on the VAS; this scale is a reliable pain assessment measure that has been validated previously
  units on a scale | 63.5 (13.9) | 68.7 (17) | 64.2 (16.2) | 65.54 (15.9)
Patient Health Questionnaire - 9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 was developed from the Primary Care Evaluation of Mental Disorders. The self-report instrument asks individuals how much they had been bothered by any of the nine problems over the prior two weeks. Items are scored from 0 (not at all) to 3 (nearly every day). Items are summed and the total score (from 0 to 27) represents the severity of depressive symptoms. 0 - 4 None-minimal None, 5 - 9 Mild, 10 - 14 Moderate, 15 - 19 Moderately Severe, 20 - 27 Severe
  units on a scale | 5.6 (3.2) | 5.9 (4.2) | 5.6 (3.5) | 5.72 (3.68)
Patient Health Questionnaire - 9 How often [Number; unit: participants] — Here we are reporting how often the patient presents symptoms? The PHQ-9 was developed from the Primary Care Evaluation of Mental Disorders. The self-report instrument asks individuals how much they had been bothered by any of the nine problems over the prior two weeks. Items are scored from 0 (not at all) to 3 (nearly every day). Items are summed and the total score (from 0 to 27) represents the severity of depressive symptoms. 0 - 4 None-minimal None, 5 - 9 Mild, 10 - 14 Moderate, 15 - 19 Moderately Severe, 20 - 27 Severe.
  participants
    Not at all | 30 | 30 | 29 | 89
    Several days | 9 | 8 | 14 | 31
    More than half the days | 2 | 4 | 0 | 6
    Nearly every day | 0 | 1 | 0 | 1
Quality of Life SF-36 [Mean (Standard Deviation); unit: units on a scale] — The SF-36 consists of 36 items addressing the patient's perception of their quality of life (QoL) in the following eight domains: physical function (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH), and one item change in health. Sub-scale scores range from 0 to 100, with 100 as the best, most positive QoL in that area and 0 is the worst. There is a total scale score, all subscales range from 0 to 100
  units on a scale
    Body pain | 38.8 (14.4) | 35.2 (14.3) | 38.5 (16.4) | 37.52 (15.2)
    Role-emotional | 66.4 (35.0) | 75.8 (38.7) | 67.2 (36.8) | 69.92 (36.89)
    Role-physical | 51.2 (40) | 51.1 (37.7) | 42.4 (37.6) | 48.21 (48.36)
    Physical functioning | 79.5 (17.8) | 72.5 (20.5) | 81.7 (11.9) | 77.91 (17.5)
    Social Function | 69.5 (22) | 68 (26.6) | 71.8 (23.6) | 69.83 (24.06)
    General health | 67.4 (18.3) | 57.3 (21.9) | 70.7 (15.4) | 65.12 (19.47)
    Mental health | 67.8 (14.2) | 65.5 (18.9) | 67.4 (17.5) | 66.93 (16.95)
    Vitality | 54.2 (13.9) | 54.7 (19.2) | 60.7 (19.3) | 56.61 (17.85)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: VAS with a score of 0-100, where 100 is the value representing the highest degree of pain and 0 the lowest. Successful treatment was defined as a reduction in pain of at least 20% of the previous score on the VAS after 4 weeks of the initial evaluation, or 14 mm on the VAS; this scale is a reliable pain assessment measure that has been validated previously
Time Frame: 4 weeks
Population: Was calculated with the software "Sample Size from Javeriana University", was taken into account an error type I of 0.05 and error type II of 0.2, number of measurements before randomization = 1, after performing scrambling = 2, correlation between measurements of 0.6, clinically important difference of 0.35, for a total number of = 45 each
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Injection + Physical Therapy | Lidocaine Injection | Physical Therapy
Number analyzed (Participants) | 41 | 43 | 43
units on a scale | 40.8 (25.3) | 44.2 (24.9) | 37.8 (21.9)

2. Secondary Outcome: PHQ 9 Function Measured With the Hand Back and Hand Mouth Maneuvers. Complications and Adverse Reactions Need for Rescue Medication
Description: The PHQ-9 was developed from the Primary Care Evaluation of Mental Disorders. The self-report instrument asks individuals how much they had been bothered by any of the nine problems over the prior two weeks. Items are scored from 0 (not at all) to 3 (nearly every day). Items are summed and the total score (from 0 to 27) represents the severity of depressive symptoms. 0 - 4 None-minimal None, 5 - 9 Mild, 10 - 14 Moderate, 15 - 19 Moderately Severe, 20 - 27 Severe
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Injection + Physical Therapy | Lidocaine Injection | Physical Therapy
Number analyzed (Participants) | 41 | 43 | 43
units on a scale | 4.33 (3.647) | 4.44 (3.03) | 4.43 (4.073)

3. Secondary Outcome: Quality of Life SF-36
Description: The SF-36 consists of 36 items addressing the patient's perception of their quality of life (QoL) in the following eight domains: physical function (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH), and one item change in health. Sub-scale scores range from 0 to 100, with 100 as the best, most positive QoL in that area and 0 is the worst. There is a total scale score, all subscales range from 0 to 100. This scale was validated in Colombia.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Injection + Physical Therapy | Lidocaine Injection | Physical Therapy
Number analyzed (Participants) | 41 | 43 | 43
units on a scale
  Changing Health | 70.0 (18.1) | 67.8 (16.05) | 60.93 (18.5)
  Body pain | 55.3 (18.4) | 51.78 (15.70) | 57.12 (20.7)
  Emotional performance | 78.2 (35.1) | 78.76 (33.24) | 85.85 (27.58)
  Physical performance | 73.1 (40.5) | 74.39 (33.3) | 73.84 (34.48)
  Physical Function | 86.8 (13.2) | 86.83 (11.55) | 82.79 (15.52)
  Social Function | 79.2 (20.7) | 78.15 (20.44) | 81.51 (22.83)
  General Health | 72.1 (16.7) | 73.54 (13.43) | 65.70 (20.16)
  Mental Health | 73.2 (16.6) | 69.95 (17.57) | 70.05 (19.82)
  Vitality | 61.3 (16) | 62.56 (17.32) | 59.88 (19.83)

4. Primary Outcome: Visual Analogue Scale
Description: as for outcome 1
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Injection + Physical Therapy | Lidocaine Injection | Physical Therapy
Number analyzed (Participants) | 41 | 43 | 43
units on a scale | 21.6 (21.8) | 28.8 (22.3) | 28.2 (23.7)

5. Secondary Outcome: PHQ 9 Function Measured With the Hand Back and Hand Mouth Maneuvers. Complications and Adverse Reactions Need for Rescue Medication
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Injection + Physical Therapy | Lidocaine Injection | Physical Therapy
Number analyzed (Participants) | 41 | 43 | 43
units on a scale | 3.98 (3.97) | 3.16 (2.81) | 4.12 (4.48)

6. Secondary Outcome: Quality of Life SF-36
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Injection + Physical Therapy | Lidocaine Injection | Physical Therapy
Number analyzed (Participants) | 41 | 43 | 43
units on a scale
  Changing Health | 70.5 (18.67) | 70.23 (17.11) | 69.76 (18.5)
  Body pain | 66.58 (20.09) | 61.19 (17.67) | 65.66 (20.9)
  Emotional performance | 83.25 (32.11) | 90.60 (21.15) | 84.13 (32.95)
  Physical performance | 81.88 (30.48) | 87.79 (22.07) | 82.5 (31.11)
  Physical Function | 87.75 (16.94) | 90 (9.06) | 89.13 (12.29)
  Social Function | 82.6 (20.99) | 83.28 (17.44) | 83.05 (20.71)
  General Health | 71.67 (17.26) | 77.44 (12.50) | 68.25 (22.37)
  Mental Health | 75.3 (16.79) | 78.95 (14.03) | 71.32 (17.86)
  Vitality | 63.38 (16.11) | 69.64 (16.17) | 61.95 (18.53)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Lidocaine Injection + Physical Therapy | Physical Therapy | Lidocaine Injection
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 4/41 | 0/43 | 3/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Injection + Physical Therapy (N=41) | Physical Therapy (N=43) | Lidocaine Injection (N=43)
Hematomas (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 2 (2) — shallow hematoma after injection of lidocaine without infectious or hemorrhagic complications.
Bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Minimal bleeding after injection of lidocaine.

LIMITATIONS AND CAVEATS:
The therapists were not the same throughout the investigation, however all were standardized to interventions; especilaistas doctors who applied the injections were different. No specific measure of patient-centered operation is used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes